CLINICAL TRIAL: NCT07356271
Title: Effects of Mouthwashes on the Oral Microbiome and Systemic Health
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Mimoza Cana-Bishop, Mrs, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: University of Plymouth
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: Oral microbiome dysbiosis
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Study Design and Appointment Structure (workflow)
  Each participant is required to attend two research appointments at either the PDSE clinic or Southside Dental Practice: first research appointment - baseline and second research appointment - follow-up (7 days after using the mouthwash). At both visits, health screening, oral checks, and sample collection are repeated. Each appointment is expected to take around one hour, based on timings from our pilot work.
  These visits are designed to collect baseline information, deliver the intervention (mouthwash or placebo), and then assess short-term changes in oral and biochemical markers following use of the mouthwash.
  1. First Research Appointment
  At this initial visit, the study is explained again in detail. Participants are given the opportunity to ask questions before providing written informed consent.
  A full oral screening is carried out.
  Oral samples (such as saliva and plaque) are collected to establish baseline m
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mouthwashes (Experimental): Population
  This study aims to recruit up to 200 participants over a period of thr years on a part-time basis. Recruitment will be carried out through three sites: (i) the University of Plymouth campus population (as successfully used in earlier studies such as Bescos et al., 2020), (ii) the Peninsula Dental School / Peninsula Dental Social Enterprise (PDSE) triage patient clinics (non-NHS clinics), and (iii) the Southside Dental Practice, a private primary care practice located in Southsea, Portsmouth.
  Sample size was calculated using G*Power software, which showed that usually 20-30 participants per group are enough, depending on whether the focus is clinical outcomes, blood markers, or microbiome changes.
  For this project, the main outcome is clinical effectiveness, measured through changes in plaque and bleeding scores.
  The PDSE clinics collectively see around 400 patients per day across their sites, providing a large and diverse pool of potential participants. In comparis
  Interventions: Drug: Use of mouthwashes
- placebo (Experimental): Population
  This study aims to recruit up to 200 participants over a period of 3 years on a part-time basis. Recruitment will be carried out through three sites: (i) the University of Plymouth campus population (as successfully used in earlier studies such as Bescos et al., 2020), (ii) the Peninsula Dental School / Peninsula Dental Social Enterprise (PDSE) triage patient clinics (non-NHS clinics), and (iii) the Southside Dental Practice, a private primary care practice located in Southsea, Portsmouth.
  Sample size was calculated using G*Power software, which showed that usually 20-30 participants per group are enough, depending on whether the focus is clinical outcomes, blood markers, or microbiome changes.
  For this project, the main outcome is clinical effectiveness, measured through changes in plaque and bleeding scores.
  The PDSE clinics collectively see around 400 patients per day across their sites, providing a large and diverse pool of potential participants. In comparis
  Interventions: Drug: Use of mouthwashes

INTERVENTIONS:
Drug: Use of mouthwashes — Population
  This study aims to recruit up to 200 participants over a period of 3 years on a part-time basis. Recruitment will be carried out through three sites: (i) the University of Plymouth campus population (as successfully used in earlier studies such as Bescos et al., 2020), (ii) the Peninsula Dental School / Peninsula Dental Social Enterprise (PDSE) triage patient clinics (non-NHS clinics), and (iii) the Southside Dental Practice, a private primary care practice located in Southsea, Portsmouth.
  Sample size was calculated using G*Power software, which showed that usually 20-30 participants per group are enough, depending on whether the focus is clinical outcomes, blood markers, or microbiome changes.
  For this project, the main outcome is clinical effectiveness, measured through changes in plaque and bleeding scores.
  The PDSE clinics collectively see around 400 patients per day across their sites, providing a large and diverse pool of potential participants. In compariso

SUMMARY:
OVERVIEW

While antimicrobial mouthwashes are proven to be clinically effective for management of certain oral microbial diseases, recent studies suggest tha, in addition to targeting bacteria responsible for gum diseases such as gingivitis and periodontitis, they may harm healthy bacteria and disturb the balance and protective role of the oral microbiome (dysbiosis).

Most findings on the oral microbiome and mouthwashes involve chlorhexidine use, demonstrating that it may induce dysbiosis and compromise the host oral microenvironment . A recent study completed in 2025 has shown that CPC mouthwash can also inhibit nitrate synthesis in the mouth. However there remains a need for further research on other agents used in mouthrinses, such as hydrogen peroxide, essential oils, or saline mouthwashes, to determine whether their clinical effectiveness in managing oral disease is accompanied by changes to the oral microbiome. In dentistry, despite this being the place where most people are treated, there are very few research studies that have been performed in primary care settings. Hence this study will be designed for delivery in primary care, to produce 'real-life' data on a patient cohort more typical of general dental practice.

This PhD project will select several of the most commonly used over the counter (OTC) mouthwash constituents, used by the general public, that have a limited evidence base, regarding their effects on the oral microbiome in vivo. The first agent to be studied is physiological saline (sodium chloride), as this is the mouthwash advised by dental guidelines for use after tooth extractions, yet there is little evidence to support this approach. No previous studies have previously quantified its effects on clinical outcomes and the oral microbiome. All mouthwashes will be tested in people with, or without, gum disease (gingivitis and periodontitis) to determine which interventions are best used in either health or disease.

DETAILED DESCRIPTION:
PROJECT AIMS

The aim of this project is to determine the role of different mouthwashes on the oral microbiome and its relationship with cardiovascular health. We will achieve this by conducting a double-blinded randomised clinical trial (pilot study) in a primary care dental setting, to investigate (i) the composition of the oral microbiome in different oral niches in periodontal health and disease, and (ii) determine how the oral microbiome is altered by the use of different mouthwashes during oral health and disease, with either physiological saline, essential oil (EOs), CPCs, hydrogen peroxide (H2O2); all versus placebo (water).

OVERVIEW

While antimicrobial mouthwashes are proven to be clinically effective for management of certain oral microbial diseases, recent studies suggest tha, in addition to targeting bacteria responsible for gum diseases such as gingivitis and periodontitis, they may harm healthy bacteria and disturb the balance and protective role of the oral microbiome (dysbiosis).

Most findings on the oral microbiome and mouthwashes involve chlorhexidine use, demonstrating that it may induce dysbiosis and compromise the host oral microenvironment. A recent study completed in 2025 has shown that CPC mouthwash can also inhibit nitrate synthesis in the mouth. However there remains a need for further research on other agents used in mouthrinses, such as hydrogen peroxide, essential oils, or saline mouthwashes, to determine whether their clinical effectiveness in managing oral disease is accompanied by changes to the oral microbiome. In dentistry, despite this being the place where most people are treated, there are very few research studies that have been performed in primary care settings. Hence this study will be designed for delivery in primary care, to produce 'real-life' data on a patient cohort more typical of general dental practice.

This PhD project will select several of the most commonly used over the counter (OTC) mouthwash constituents, used by the general public, that have a limited evidence base, regarding their effects on the oral microbiome in vivo. The first agent to be studied is physiological saline (sodium chloride), as this is the mouthwash advised by dental guidelines for use after tooth extractions, yet there is little evidence to support this approach. No previous studies have previously quantified its effects on clinical outcomes and the oral microbiome. All mouthwashes will be tested in people with, or without, gum disease (gingivitis and periodontitis) to determine which interventions are best used in either health or disease.

BACKGROUND

1. Introduction to the Oral Microbiome

   The oral cavity is one of the most ecologically diverse habitats in the human body, hosting hundreds of microorganisms such as bacteria, archaea, fungi, protozoa, and viruses that coexist within biofilms on both soft and hard oral tissues. The oral microbiome is now understood to not be a passive community but is rather a highly dynamic, interactive, immunologically and metabolically active system, not just orally but both in oral and systemic health Historically, the study of oral microorganisms was restricted by culture-based techniques. While these methods were important in identifying cariogenic species such as Streptococcus mutans and periodontal pathogens such as Porphyromonas gingivalis, they dramatically underestimated microbial diversity because only a minority of oral species can be cultured under laboratory conditions. With the introduction of 16S ribosomal RNA (rRNA) gene sequencing and later shotgun metagenomics, the true complexity of the oral microbiome was revealed. These methods identified more than 700 bacterial taxa, along with a wide variety of fungi (e.g., Candida spp.), viruses (including bacteriophages), and protozoa.

   The oral microbiome is not the same everywhere in the mouth; it is site-specific. Different areas, such as saliva, plaque, the tongue and gingival crevicular fluid (GCF), each host their own unique mix of microorganisms. These communities are shaped by factors like the immune system, pH levels, oxygen, and available nutrients. Because of this, oral health and disease cannot be fully understood by studying saliva alone; samples from multiple sites are needed to capture the full picture. In each of these niches, in oral health these populations are diverse, whereas in oral disease, the oral microbiome becomes less diverse and pathogenic species predominate. For example, in supra-gingival plaque, one NGS study found higher abundance of bacteria associated with gingivitis, such as Fusobacterium, Treponema and Campylobacter and lower abundance of bacteria associated with oral and cardiovascular health, such as Neisseria, Actinomyces, and Rothia.
2. Dysbiosis of oral microbiome

   Dysbiosis is a disruption of microbial balance leading to a dominance of pathogenic species and loss of symbiosis. In the oral cavity, dysbiosis underlies the host response and clinical outcomes for most prevalent dental diseases, including dental caries, gingivitis and periodontal diseases.

   2.1. Dysbiosis of oral microbiome in oral disease

   Dental caries (tooth decay) is mainly caused by Streptococcus mutans. This bacterium feeds on sugars from food and produces acid, which demineralises the enamel and dentine. It often hides in the pits and grooves of teeth and forms sticky biofilms. When S. mutans combines with fungi like Candida albicans, the biofilms become even stronger and more harmful. This partnership is especially linked to early childhood caries. Because tooth decay is still the most common disease worldwide, researchers are exploring new treatments, such as probiotics that add "good bacteria" and medicines that can target S. mutans more directly.

   Plaque results in the inflammation of gingival tissue and gingivitis in some forms are estimated to affect up to 90% of the world's population at one time or another. It is reversible, but if left untreated can be a precursor to irreversible periodontal diseases. In humans, gingivitis typically arises in response to communities of bacteria (dental plaque) attached to the surface of teeth (supra-gingivally) in people with poor oral hygiene. Clinically, gingival inflammation is seen as bleeding when the gingival is probed, as well as redness and swelling of the gingival marginal tissues, without any signs of periodontal attachment loss. Being reversible, gingivitis is a condition that can be managed effectively with therapy and improved oral hygiene. However, if left untreated, it can progress to periodontitis

   Gingivitis can be linked to bacteria such as Leptotrichia buccalis and Prevotella species, as these are found to predominate in the plaque of people with gingivitis ) These bacteria can trigger the body's immune system to release inflammatory molecules, causing redness, swelling, and bleeding of the gums. While Leptotrichia is normally harmless, it may play a part in gum inflammation when conditions in the mouth change. Prevotella species are more directly involved, as they are often found in higher numbers when gums become inflamed.

   Periodontitis manifests clinically with bleeding on probing (BOP) from deeper periodontal pockets and eventually tooth mobility and loss due to the irreversible destruction of alveolar bone, which holds teeth in place. Pockets are first created due to localised host inflammation and swelling in response to pathogenic Gram-negative bacteria present in plaque below the gumline (sub-gingival), such as Porphyromonas gingivalis, Fusobacterium, Treponema and Tannerella species . The inflammatory mediators that are released into the pocket in response to this infection, also destroy bone, which further deepens the pockets and makes oral hygiene even more challenging.

   Two of the most important bacteria that predominate in the oral microbiome of people with periodontal disease include Porphyromonas gingivalis and Fusobacterium nucleatum.

   P. gingivalis is a Gram-negative, anaerobic bacterium that grows without oxygen' This bacterium thrives when the mouth's microbial balance, or microbiome, is disturbed. In these conditions, it triggers inflammation, which contributes to the development of gum disease. One of the reasons P. gingivalis is so harmful is its ability to invade human cells, resist some antibiotics, and use thin, hair-like structures called fimbriae to attach to and enter host cells. Beyond gum disease, it is also linked to oral and digestive cancers. It encourages cells to grow while avoiding normal cell death, blocks tumour-suppressor proteins such as p53, and triggers cell changes (epithelial-mesenchymal transition, EMT) that allow cancer to spread. Because of these factors, P. gingivalis is considered a dangerous pathogen that not only causes periodontal disease but also increases the risk of oral cancer.

   F. nucleatum is another Gram-negative, anaerobic bacterium that is very common in the mouth. While it was once thought to be harmless, it is now recognised as an important disease-causing organism. It has also been found outside the oral cavity in several conditions, including bowel disease, colorectal cancer, Crohn's disease, arthritis, meningitis, appendicitis, and pregnancy complications. Within the mouth, F. nucleatum plays a key role in dental biofilms, acting as a bridge that connects different bacterial species. It uses proteins such as FadA and Fap2 to stick to human cells, provoke inflammation, and promote tumor growth. The bacterium stimulates immune signals like IL-6, IL-8, IL-17, and TNF-α. While these signals support healing in healthy conditions, in disease they contribute to DNA damage and cancer. F. nucleatum is also capable of resisting antibiotics and reducing the effectiveness of certain cancer treatments. It is often found alongside P. gingivalis in oral cancers, and together these bacteria strongly enhance pathways that promote cancer growth.

   2.2. Treatment of oral disease

   At the dentist, gingivitis is managed with improved oral hygiene instruction; OHI (tooth brushing and interdental cleaning); dentists and dental hygiene therapists promote at home oral hygiene regimens, as the most important factor for the stabilisation of the disease. In periodontitis, OHI is accompanied by non-surgical therapy performed within the dental practice, usually every 3 months (supra- and sub-gingival scaling with ultrasonic or hand scalers known as PMPR), to reduce bacterial load within the periodontium. Indeed, the diversity of the oral microbiome increases after PMPR, and PMPR leads to immediate reduction in periodontal inflammation (Johnston et al,2023). This is because bacterial load is reduced, such that the structure of the plaque is less favourable for many of the pathogenic anaerobic bacteria associated with oral disease. Despite this, many patients do not maintain improvements in periodontal health after OHI and PMPR, and new adjunctive measures such as mouthwash are often sought, for example in patients with impaired dexterity, and other mental or physical health conditions which can impair engagement.
3. Links Between Oral Microbiome and Systemic Health

   Importantly, dysbiosis is not just the presence of pathogens but an imbalance where protective microorganisms decline and pathogenic taxa dominate. In the past decade, the interest in the oral microbiome by researchers has grown, as an important link in systemic health. There is a growing body of evidence linking periodontal disease and systemic diseases, such as diabetes, cardiovascular disease, Alzheimer's. The evidence for cardiovascular disease is some of the most compelling and there are several systematic reviews and meta-analysis that report on the association between periodontal disease and cardiovascular disease, including hypertension. The systematic review by Munoz-Aguilera found a clear link between periodontitis and hypertension. Patients with moderate to severe gum disease were about 20% more likely to have high blood pressure than those without, and the risk increased with disease severity. On average, people with periodontitis had higher blood pressure readings; around 4.5 mmHg systolic and 2 mmHg diastolic. These findings suggest that periodontitis may be a modifiable risk factor for hypertension. The review also considered possible mechanisms. Periodontitis can drive systemic inflammation, releasing molecules like CRP, IL-6, and TNF-α that impair blood vessel function. Oral bacteria such as Porphyromonas gingivalis may also directly affect vascular health and blood pressure. Overall, the evidence indicates that gum disease and hypertension are closely linked, and periodontal therapy could play a role in reducing cardiovascular risk.

   There are several different mechanisms that have been proposed for this relationship: (1) systemic inflammation due to cytokines released into the bloodstream during bacterial dysbiosis, (2) bacteraemia (pathogenic oral bacteria entering the bloodstream), (3) the oral bacterial enterosalivary pathway (with systemic nitric oxide [NO] release), and (4) genetic susceptibility . Genetic factors, pre-existing disease and the host response also play a part in terms of the amount of inflammation and clinical outcomes observed in response to oral microbiome dysbiosis. However, this study will focus on the salivary-entero nitrate reducing pathway involving nitric oxide, as our previous studies have demonstrated that this is affected by mouthwashes

   3.1 Cardiovascular Health

   In health there are bacteria on the dorsum of the tongue (and thus saliva), that convert nitrate in food to nitrite, which is swallowed and converted into nitric oxide (NO) in the gut wall to maintain a lower blood pressure. Nitrates and nitrites widely exist in soil, water, and plants. Humans get their nitrates through food, mainly through green vegetables. These dietary nitrates are stable but when in contact with symbiotic bacteria in the oral cavity and stomach, they get converted to nitrite and nitric oxide (NO). NO is the metabolic product of dietary nitrate and plays an important role in protecting cardiovascular system and gastric mucosa. Via this mechanism therefore, nitrate-reducing oral bacteria can module blood pressure.

   In the oral cavity these nitrate-nitrite reducing bacteria tend to be in the deep crypts of the posterior part of the tongue , but can also be identified in saliva . Those species in the mouth that are nitrate reducing can be broadly categorised into two groups: strict anaerobes (Veillonella atypica and Veillonella dispar) and facultative anaerobes (Actinomyces odontolyticus and Rothia mucilaginosa). Veillonella species have been identified as the primary nitrate reducers in the tongue and play a significant role in nitrate reduction. Recent research utilising 16S rRNA has revealed a higher prevalence of Prevotella, Neisseria and Haemophilus on the posterior surface of tongue compared with Actinomyces . The presence of sufficient nitrate reducing bacteria when exposed to dietary nitrates, therefore, play an important role in prevention of myocardial infarctions, hypertension, and acute stress, due to its role as a biological reservoir for NO in hypoxia or acidic conditions. A moderate consumption of nitrate rich fruits and vegetables such as beetroot, spinach, lettuce, radish and celery, therefore, is a low-cost way of contribution to cardiovascular health in part via the oral microbiome .
4. Mouthwashes as Modifiers of the Oral Microbiome

4.1. Clinical effectiveness

A huge variety of mouthwashes are available over the counter and can be either chemical or natural. Some of the most commonly used antimicrobial mouthwashes include chlorhexidine (CHX), hydrogen peroxide (H2O2), cetylpyridinium chloride (CPC), povidone iodine (PVP-I), and essential oils (EO) . These mouthwashes are used because they are clinically effective in terms of reducing plaque and bleeding, and in turn gingivitis . They also have a small degree of clinical effectiveness, particularly chlorhexidine, at reducing pocket depths when used adjunctively alongside OHI and PMPR . Thus, they are widely used by patients as an over-the counter (OTC) treatment to address problems such as bleeding gums and bad breath (halitosis). However, they are also integrated into the daily oral hygiene routines of healthy individuals, and thus it is important to evaluate whether there is oral dysbiosis in this group, as mouthwashes should ideally be used only when benefits outweigh risks

4.2. Mechanism of action and clinical effectiveness

4.2.1. Chlorhexidine digluconate

Chlorhexidine has been used in medicine and dentistry since 1950, being found in mouthwashes since1970. It has been used as an effective antiseptic agent for 'killing' both gram positive and negative bacteria, fungi, and certain viruses. A study by Rius-Salvador et al., 2024 indicated that Chlorhexidine can decrease the infectivity of both the Influenza A virus and the Respiratory Syncytial virus in vitro.

Chlorhexidine is a bacteriostatic at lower concentrations of 0.02%-0.06%, and bactericidal at the higher concentration of 0.12%. Chlorhexidine is used in dentistry as an antiseptic mouthwash at 0.12%-0.2% and surface disinfectant at 0.2% for this reason. Chlorhexidine is a positively charged cationic bisbiguanide that can be adsorbed to a variety of negatively charged sites, including mucous membranes, salivary pellicle on teeth, as well as several components of the biofilm on the tooth surfaces, e.g., bacteria, extracellular polysaccharides, and glycoproteins. In vitro studies have showed that, at concentrations lower than used clinically, chlorhexidine causes destruction to the cell membrane and in turn and low molecular weight molecules escape from the microorganisms. On the other hand, a higher concentration of chlorhexidine can cause precipitation and coagulation of the proteins in the cytoplasm of the exposed microbes. These properties interfere with biofilm formation and prevent bacterial growth .

One of the systematic reviews confirmed that the daily chlorhexidine mouthwash (used alongside brushing/flossing) greatly reduces dental plaque over 4-6 weeks, and this effect is maintained up to 6 months. The same study also confirmed a high- certainty evidence that chlorhexidine reduces gingivitis in people with mild gum inflammation, with consistent improvements seen both short- and long-term. In periodontal disease, studies also prove that it is clinically effectively at reducing periodontal pockets when used adjunctively. A meta-analysis confirmed that adjunctive use of chlorhexidine mouth rinse with mechanical scale and root planning (SPR) resulted in slightly greater probing depth reduction than did SRP alone.

Chlorhexidine also reduces Streptococcus mutans levels, suggesting possible benefits in preventing tooth decay, but more long-term, high-quality studies are needed to confirm this. In terms of other oral health benefits, a 2019 systematic review by found low certainty evidence that chlorhexidine mouthwash may help reduce bacteria that cause halitosis. A 2022 Cochrane review found moderate-certainty evidence that chlorhexidine rinses before and after tooth extraction lower the risk of dry socket.

Beyond dentistry, a 2020 Cochrane review suggested chlorhexidine may lower the risk of ventilator-associated pneumonia in critically ill patients (low-certainty evidence). During COVID-19, interest in pre-procedural mouthwashes grew, but current evidence is insufficient to confirm benefits for patient outcomes or healthcare worker safety.

4.2.2. Essential oils (EO)

It is difficult to find antimicrobial data for essential oils alone, in terms of the mechanisms and clinical effectiveness when they are used as a mouthwash, but the base for EO mouthwashes such as in ListerineTM, traditionally includes thymol, methyl salicylate and eucalyptol. Traditionally, the mechanism of action of essential oils is thought to be based on disruption of cytoplasmic membranes and inhibition of bacterial enzymes, however, despite many studies describing the antimicrobial activities of essential oils, herbal extracts, or their active components, there remains a lack of evidence on their mechanisms of action . ListerineTM can reduce plaque and bleeding scores and therefore reduce clinical signs of gingivitis . It is also recommended adjunctively for periodontal disease however, ListerineTM contains alcohol (plus CPCs in some formulations), which complicates knowledge and understanding of the true mechanisms on EOs in vivo. Thus, further clinical studies are required to elucidate the clinical effects of EOs alone. Alcohol may also affect the oral microenvironment, and whilst unfounded, regarding the risk of alcohol mouthwashes causing cancer there are still some concerns about the suitability of daily use of alcohol mouthwashes by pregnant women, those with alcohol dependency and in patients with mucosal injuries. Consequently, the alcohol free EO mouthwashes have been introduced by ListerineTM and others .

4.2.3 Hydrogen peroxide (H2O2)

H2O2 has found its application in dentistry for more than 70 years either in combination with salt or in its pure form. H2O2 has been shown to possess a wide spectrum of antimicrobial activity because it is active against bacteria, yeasts, fungi, viruses, and spores, however these positive outcomes are observed with concentrations greater than 1% . H2O2 is a bleaching agent with strong oxidising action that releases free radicals and disrupts the lipid component of microbial cell wall . In addition, H2O2 produces foam when in contact with human tissue, releasing water and oxygen which is believed to contribute to the destruction of anaerobic bacterial species.

A 5% concentration of H2O2 causes soft tissue damage, therefore it is used in dentistry as antiseptic mouthwash at concentrations of 1.5%-3.0% . A systematic review done in 2011 showed that H2O2 mouthwashes do not consistently prevent plaque accumulation when used as a short-term mono-therapy. When used as a long-term adjunct to daily oral hygiene however, one study indicated that oxygenating mouthwashes reduce gingival redness. This systematic review was limited by what was available in the existing dental literature and found that only one study that had an evaluation period of more than 4-weeks. Therefore, the outcome of this review with respect to levels of gingival inflammations was based on a single experiment with an estimated low risk of bias. Clearly, this is not sufficient evidence to draw any conclusions on, regarding the long-term effects of H2O2 on plaque levels.

4.2.4.Cetylpyridinium chloride (CPC)

CPCs are found in many commercially available OTC mouthwashes, and are classified as quaternary ammonium compounds (QACs) that are antibacterial because they react with lipids and proteins of cell membrane, causing leakage of low molecule components. CPCs can also cause the release cytolytic enzymes, leading to the lysis of bacterial cells . It is worth noting that QACs are also commonly used in various surface spray disinfectants, so have other uses within the dental surgery . They are used in mouthwashes at varying concentrations (0.045%-0.1%). The results of a clinical trial demonstrated that the use of a 0.07% CPC mouth rinse was significantly more effective in reducing plaque scores than the use of the Vehicle Control (VC) mouth rinse. However, there were no significant differences between the CPC and VC groups, with respect to bleeding scores observed at 6 months. CPC's may also be effective in reducing plaque and the levels of anaerobic species of bacteria in plaque and saliva , however, evidence from in vivo studies remains limited . Similar to EOs, CPCs are usually used in combination with other effective antibacterial agents, including CHX and alcohol, as well as fluoride. Thus, further studies are required investigating the antibacterial effects of CPCs alone, rather than commercially available products whose formulations are very complex and change over time.

4.2.5 Saline rinses

Saline refers to an isotonic solution containing sodium chloride (NaCl), and water, usually of concentrations of 0.09% when referred to a 'physiological' saline. However, at higher concentrations it may be antibacterial.The literature suggests that 1.4-1.7% is the appropriate concentration to use in saline mouth rinses but there is some uncertainty about this in clinical dentistry, and hence determining a clinically relevant concentration also forms part of this thesis. Although, it is arguably less potent as an antimicrobial agent than some of the chemical agents discussed thus far, it has been recognised for its mild antiseptic properties for centuries and is still advised by dental practitioners on a daily basis for managing oral infections . It is difficult therefore to understand, the lack of evidence-base surrounding the appropriate dose and frequency of saline use in dentistry.

Based on what evidence does exist, it has been suggested that saltwater or saline mouth rinses can reduce plaque scores and the colony counts in saliva of bacteria in vitro, such as S mutans, L acidophilus, A actinomycetemcomitans, and P gingivalis . Saline also reduces the pH within the oral cavity in vivo, and may cause bacteria to lose water due to osmosis; thus, it makes sense that saltwater reduces the growth of unwanted oral bacteria. As mentioned, dental practitioners often suggest saltwater rinses for postoperative care after oral surgery, but there is little evidence to support this recommendation, and hence the clinical effectiveness and antibacterial mechanisms of saline mouth rises requires further investigation

Saline is also commonly regarded as being beneficial for reducing gingival inflammation and facilitating the healing of oral ulcerative lesions. An in vitro study performed by Huynh et al., in 2016 used human gingival fibroblasts (hGFs) cultured in growth medium already containing a small amount of NaCl (about 0.4%). In this study cells were therefore exposed to slightly higher dosages of NaCl than in saline mouth rinses, showing that 1.8% NaCl was the most effective concentration at stimulating hGF cell migration, altering the organisation of cytoskeletal molecules (FAK and F-actin), and enhancing extracellular matrix gene expression (COL1 and Fn). These data provided the first scientific evidence to support the application of salt solution as mouthrinse in conjunction with routine oral care to promote oral wound healing. Saline rinses are thus recommended post-extraction for wound healing as part of national guidelines .They have further been shown to alleviate xerostomia, reduce halitosis, and significantly lower bacterial load within the oral cavity , yet evidence on their clinical effectiveness due to an antibacterial effect in vivo is virtually absent.

4.2.6. Fluoride (mouthwashes)

Fluoride is widely used, and it's found in various oral products such as toothpaste mouthwash and gels. Mouthwashes are particularly favoured by the public due to their easy use, and recommendations in current guidelines

Fluoride mouthwashes have been widely recommended for maintaining oral health, especially in the prevention of dental caries. Sodium fluoride is the most common active ingredient. Fluoride concentration in these rinses varies: OTC products usually contain about 200-1000 ppm, while prescription formulations may contain several thousand ppm. Typically, OTC mouthwashes are intended for daily use, whereas prescription-strength rinses are used less frequently. Although fluoride is known to have some antiplaque activity, there is limited direct evidence on its effectiveness in reducing plaque levels or in managing gingivitis and periodontal disease when used as a mouthwash .A 2016 undertook a systematic review, finding that supervised regular use of fluoride mouthrinse by children and adolescents was associated with a large reduction in caries compared with control groups, on average by 27%, but there was no such similar study in adults

There is no evidence for effects of mouth rinses with fluoride on dental plaque accumulation, gingivitis development or periodontal disease in vivo. In vitro, sodium fluoride mouthwash had little effect on P gingivalis, P intermedia, F nucleatum, and A actinomycetemcomitans; using ex vivo cultures of bacteria from the tongue . Thus, given the widespread use of fluoride-containing mouthwashes, there is much work to be done in terms of quantifying the clinical effectiveness of fluoride on periodontal health in vivo and the antimicrobial mechanisms associated with this. Perhaps the known anti-caries benefits of fluoride outweigh the need to know this clinically, but the marketing of these fluoride-containing mouthwashes does often pertain to improving gum health.

4.2.7. Alternatives: Herbal and Probiotic Rinses.

There is growing consumer demand for "natural" products, and within mouthwashes this has incited interest in alternatives such as:

Coconut oil (pulling)

Seaweed

Propolis

Probiotic rinses

ELIGIBILITY:
* Inclusion & Exclusion

All individuals aged 18 years and older will be eligible to take part in this study. Exclusion will apply to individuals who:

Are current smokers, due to the well-documented impact of smoking on oral and systemic health.

Have a known diagnosis of hypertension, diabetes, or cancer, as these systemic conditions may influence oral microbiome and inflammatory responses.

Have taken a course of antibiotics within the last three months, since antibiotics are known to disrupt microbial balance and may confound the interpretation of oral microbiome data.

Report allergies to essential oils or to milk proteins, as these ingredients may be present in the study mouthwash and could trigger adverse reactions.

In addition, participants who have never previously used a mouthwash will be excluded. This is a precautionary measure designed to avoid even the minimal possibility of adverse responses, since prior tolerance to similar products suggests a reduced risk of sensitivity Since their introduction in the 1970s, chlorhexidine-containing mouthwashes have only rarely been linked to immune-mediated reactions. Reported cases include type IV hypersensitivity after mouthwash use, type I hypersensitivity following treatment with chlorhexidine dental gel or disinfection of a lip injury, and urticarial skin lesions after rinsing with chlorhexidine. More seriously, two recent cases in the UK reported fatal anaphylaxis linked to the use of chlorhexidine mouthwash after tooth extraction (Pemberton 2016).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
effect of mouthwashes on oral microbiome | three years
  EXPECTED OUTCOMES / DELIVERABLES
  One of the main expected outcomes of this study is to provide clear evidence on the clinical effectiveness of commonly used mouthwashes and their effect on oral microbiome and cardiovascular health. It is anticipated that some mouthwashes will significantly reduce dental plaque and bleeding on probing when compared with placebo. Demonstrating these effects will help confirm which products can genuinely support daily oral hygiene and clinical treatment of gum conditions, alongside either beneficial or no effects on the oral microbiome, such that their beneficial effects do not outweigh the risks.
  In participants with good oral health, we thus expect that effective mouthwashes will not only reduce plaque but also maintain a balanced oral microbiome. This means that mouthwashes should support microbiome health, without causing dysbiosis or loss of diversity.
  In participants with gingivitis or periodontal disease, the expectation is that mouthwash

SECONDARY OUTCOMES:
effect of mouthwashes on cardiovascular health | three years
  EXPECTED OUTCOMES / DELIVERABLES
  One of the main expected outcomes of this study is to provide clear evidence on the clinical effectiveness of commonly used mouthwashes and their effect on oral microbiome and cardiovascular health. It is anticipated that some mouthwashes will significantly reduce dental plaque and bleeding on probing when compared with placebo. Demonstrating these effects will help confirm which products can genuinely support daily oral hygiene and clinical treatment of gum conditions, alongside either beneficial or no effects on the oral microbiome, such that their beneficial effects do not outweigh the risks.
  In participants with good oral health, we thus expect that effective mouthwashes will not only reduce plaque but also maintain a balanced oral microbiome. This means that mouthwashes should support microbiome health, without causing dysbiosis or loss of diversity.
  In participants with gingivitis or periodontal disease, the expectation is that mouthwash

CONTACTS AND LOCATIONS:
Overall Officials: zoe Brookes, PhD, Study Director — University of Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] References Al-Maweri, S. A., et al. (2025). "The association between the oral microbiome and hypertension: a systematic review." Journal of oral microbiology 17(1): 2459919. Alrashdan, M. S., et al. (2023). "The Effects of Antimicrobial Mouthwashes on Systemic Disease: What Is the Evidence?" International dental journal 73: S82-S88 Aravinth, V., et al. "Comparative evaluation of saltwater rinse with chlorhexidine against oral microbes: a school-based randomized controlled trial " Indian Soc Pedod Prev Dent, 35 (4) (2017), pp. 319-326 Bescos, R., et al. "The comparative effect of propolis and chlorhexidine mouthwash on oral nitrite-producing bacteria and blood pressure regulation." Bescos, R., et al. (2020). "Effects of Chlorhexidine mouthwash on the oral microbiome." Sci Rep 10(1): 5254-5254. Bondonno, C. P., et al. (2015). "Antibacterial Mouthwash Blunts Oral Nitrate Reduction and Increases Blood Pressure in Treated Hypertensive Men and Women." Am J Hypertens 28(5): 572-575. Brookes, Z., et al. (2023). "Antimicrobial Mouthwashes: An Overview of Mechanisms-What Do We Still Need to Know?" International dental journal. Brookes, Z., et al. (2023). "Mouthwash Effects on the Oral Microbiome: Are They Good, Bad, or Balanced?" International dental journal. Burcham, Z. M., et al. (2020). "Patterns of Oral Microbiota Diversity in Adults and Children: A Crowdsourced Population Study." Scientific reports 10(1): 2133. Burton, J. P., et al. (2006). "preliminary study of the effect of probiotic Streptococcus salivarius K12 on oral malodour parameters." Journal of Applied Microbiology 100(4): 754-764. Casarin, M., et al. (2023). "Effect of mouthwashes on gingival healing after surgical procedures: A systematic review." European Journal of Oral Sciences 131(3): e12931-n/a. Caselli, E., et al. (2020). "Defining the oral microbiome by whole-genome sequencing and resistome analysis: the complexity of the healthy picture." BMC Microbiol 20(1): 120-120
- See also: Library of Plymouth university that covers the main databases — https://primo.plymouth.ac.uk/discovery/search?vid=44PLY_INST:VU_PLY